CLINICAL TRIAL: NCT05988073
Title: A Multicenter Prospective Longitudinal Study of Clinical Outcomes, Disease Course, Health-Related Quality of Life, and Health Care Resource Utilization in Adult Patients With Multifocal Motor Neuropathy
Brief Title: A Prospective Longitudinal Study in Adults With Multifocal Motor Neuropathy
Acronym: iMMersioN
Status: Active, not recruiting | Type: Observational
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Other Study IDs: ARGX-117-2202
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2025-06-20 (Actual); Status verified 2025-06

CONDITIONS: Multifocal Motor Neuropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This prospective longitudinal study will follow participants with Multifocal Motor Neuropathy over time and collect data on their clinical outcomes, quality of life, and use of health care resources. Participants will follow their regular visit schedule with their treating physician, except for an optional second visit occurring 7 to 14 days after the start of the study to collect biomarker data. No IMP will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Is at least the local legal age of consent for clinical studies when signing the ICF
* Is capable of providing signed informed consent and complying with protocol requirements
* Has an existing or new diagnosis of MMN made by a neuromuscular specialist or neurologist

Exclusion Criteria:

* Is currently participating in any clinical study with an IMP
* Has other medical conditions that could affect the assessment of MMN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with MMN receiving standard of care at their treating physician.
Sampling Method: Probability Sample
Enrollment: 413 (Actual)
Dates: Start 2023-11-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To characterize MMN patient profiles for participants | up to 37 months
To assess the MMN disease management and disease course | up to 37 months
To assess outcome measures specific to MMN disease and their evolution over time | up to 37 months
To estimate the burden of MMN on participants' quality of life | up to 37 months
To estimate the economic burden for participants with MMN | up to 37 months
To collect data on relevant disease biomarkers | up to 37 months

CONTACTS AND LOCATIONS:
Locations (113):
- United States (24):
  - Neuromuscular Clinical and Research Center, Phoenix, Arizona
  - HonorHealth Neurology - Bob Bove Neuroscience Institute, Scottsdale, Arizona
  - UCI Health - ALS and Neuromuscular Center, Orange, California
  - Stanford Medicine Health Care - Stanford Neuroscience Health Center, Palo Alto, California
  - The Neurology Group, Pomona, California
  - Eisenhower Health - Rancho Mirage Medical Center, Rancho Mirage, California
  - UC Davis Health - Lawrence J. Ellison Ambulatory Care Center, Sacramento, California
  - UCSF Health - UCSF Medical Center, San Francisco, California
  - University of Colorado - Anschutz Medical Campus, Aurora, Colorado
  - YaleNewHavenHealth - Yale New Haven Hospital, New Haven, Connecticut
  - MedStar Health - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Medsol Clinical Research Center Inc, Port Charlotte, Florida
  - D&H National Research Centers - Tamarac Research Center, Tamarac, Florida
  - Hospital Sisters Health System (HSHS) - St Elizabeth's Hospital, O'Fallon, Illinois
  - The University of Kansas Health System - Landon Center on Aging, Kansas City, Kansas
  - Rutgers University - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Columbia University Irving Medical Center - Neurological Institute of New York, New York, New York
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Ohio State University Wexner Medical Center - Ohio State Martha Morehouse Outpatient Care, Columbus, Ohio
  - Oregon Health and Science University (OHSU) Hospital - Marquam Hill Campus, Portland, Oregon
  - Penn Medicine - Penn Medicine University City, Philadelphia, Pennsylvania
  - Penn Medicine - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Northwest Houston Neurology - Cypress, Cypress, Texas
- Australia (3):
  - Royal Melbourne Hospital, Parkville
  - Gold Coast University Hospital, Southport
  - Princess Alexandra Hospital, Woolloongabba
- Allgemeines Krankenhaus der Stadt Wien (AKH Wien), Vienna, Austria
- Belgium (7):
  - Hopital Erasme, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - Universitair Ziekenhuis Brussel, Jette
  - Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven
  - L'hopital de la Citadelle - Site Citadelle, Liège
  - Cliniques Universitaires Saint-Luc, Woluwe-Saint-Lambert
- Bulgaria (4):
  - Multiprofile Hospital for Active Treatment - Uni Hospital OOD, Panagyurishte
  - Medical Center Medconsult Pleven OOD, Pleven
  - Military Medical Academy - Military Hospital for Active Treatment Pleven, Pleven
  - University Multiprofile Hospital for Active Treatment and Emergency Medicine N. I. Pirogov, Sofia
- Canada (5):
  - London Health Sciences Centre - University Hospital, London
  - Centre Hospitalier de l'Universite de Montreal, Montreal
  - McGill University Health Centre - The Neuro (Montreal Neurological Institute-Hospital), Montreal
  - CHU de Quebec - Hopital de L'enfant Jesus, Québec
  - University of Saskatchewan - University of Saskatchewan College of Medicine, Saskatoon
- China (3):
  - Xiangya Hospital of Central South University, Changsha
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Huashan Hospital of Fudan University, Shanghai
- Czechia (2):
  - Fakultni nemocnice Brno - Areal Bohunice, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
- Denmark (2):
  - Aarhus Universitetshospital, Aarhus
  - Rigshospitalet - Blegdamsvej, Copenhagen
- France (11):
  - CHU Angers, Angers
  - CHU de Bordeaux - Hôpital Pellegrin, Bordeaux
  - CHU Brest - Hopital La Cavale Blanche, Brest
  - Hospices Civils de Lyon (HCL) - Hopital Pierre Wertheimer, Bron
  - Assistance Publique Hopitaux de Paris (AP-HP) - Hopital Bicetre, Le Kremlin-Bicêtre
  - CHU Lille - Hopital Salengro, Lille
  - CHU de Limoges - CHU Dupuytren 1, Limoges
  - AP-HM - CHU Timone, Marseille
  - CHU de Nantes - Hotel Dieu, Nantes
  - CHU de Nice - Hopital Pasteur, Nice
  - Assistance Publique Hopitaux de Paris (AP-HP) - Hopital Pitie-Salpetriere, Paris
- Germany (5):
  - Universitatsklinikum Essen, Essen
  - Universitatsklinikum Giessen und Marburg - Campus Giessen, Giessen
  - Medizinische Hochschule Hannover, Hanover
  - St. Josefs- Krankenhaus Potsdam- Sanssouci, Potsdam
  - Universitatsklinikum Wurzburg, Würzburg
- Italy (10):
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Fondazione Serena Onlus - NeMO Brescia, Gussago
  - Azienda Ospedaliera Universitaria Gaetano Martino, Messina
  - Universita degli Studi del Piemonte Orientale Amedeo Avogadro - Scuola di Medicina, Novara
  - Azienda Ospedaliero-Universitaria San Luigi Gonzaga, Orbassano
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo
  - Istituto Neurologico Nazionale a Carattere Scientifico IRCCS, Pavia
  - Azienda Ospedaliero Universitaria Pisana - Ospedale Santa Chiara, Pisa
  - Azienda Ospedaliero Universitaria Sant'Andrea, Roma
  - Fondazione PTV Policlinico Tor Vergata, Roma
- Japan (3):
  - Teikyo University Hospital, Itabashi-ku
  - National Center of Neurology and Psychiatry, Kodaira-shi
  - Dokkyo Medical University Hospital, Mibu
- Latvia (2):
  - Riga East Clinical University Hospital, Riga
  - Pauls Stradins Clinical University Hospital, Riga
- Poland (9):
  - Medicover Integrated Clinical Services (MICS) - Centrum Medyczne Bydgoszcz, Bydgoszcz
  - Wielospecjalistyczna Poradnia Lekarska Synapsis, Katowice
  - Specjalistyczne Gabinety Sp. z o.o., Krakow
  - Michalski i Partnerzy Lekarze Spolka Partnerska, Krakow
  - SP ZOZ Szpital Uniwersytecki w Krakowie, Krakow
  - CLINIREM Sp z o.o., Lublin
  - Rejdak Konrad Indywidualna Praktyka Lekarska, Lublin
  - Centrum Medyczne Hope Clinic, Lublin
  - ETG Network - ETG Neuroscience, Warsaw
- Spitalul Clinic Judetean de Urgenta Sf. Apostol Andrei, Constanța, Romania
- Serbia (2):
  - Univerzitetski klinicki centar Srbije, Belgrade
  - Univerzitetski klinicki centar Kragujevac, Kragujevac
- Spain (8):
  - Hospital General Universitario Dr. Balmis, Alicante
  - Hospital Universitari Germans Trias i Pujol (HUGTP), Badalona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario de Basurto, Bilbao
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario de Navarra, Pamplona
  - Hospital Universitario de Donostia, San Sebastián
- Sweden (2):
  - Sahlgrenska Universitetssjukhuset - MS - mottagning Sahlgrenska, Gothenburg
  - Karolinska Universitetssjukhuset - Huddinge, Huddinge
- United Kingdom (9):
  - North Bristol NHS Trust - Southmead Hospital Bristol, Bristol
  - Lancashire Teaching Hospitals NHS Foundation Trust - Royal Preston Hospital, Fulwood
  - NHS Great Glasgow and Clyde - Queen Elizabeth University Hospital, Glasgow
  - Nottingham University Hospitals NHS Trust - Queen's Medical Centre, Nottingham
  - Oxford University Hospitals NHS Foundation Trust - John Radcliffe Hospital, Oxford
  - Northern Care Allicance NHS Foundation Trust - Salford Royal, Salford
  - Sheffield Teaching Hospitals NHS Foundation Trust - Royal Hallamshire Hospital, Sheffield
  - Somerset NHS Foundation Trust - Musgrove Park Hospital, Taunton
  - Royal Cornwall Hospitals NHS Trust - Royal Cornwall Hospital, Truro

IPD SHARING:
Plan to Share IPD: No